CLINICAL TRIAL: NCT03559270
Title: A Multicenter, Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Baricitinib (LY3009104) in Participants With Moderate to Severe Atopic Dermatitis
Acronym: BREEZE-AD6
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to lack of alignment during regulatory negotiations.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17064; I4V-MC-JAIX (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo/Baricitinib 2-milligram (mg) (Experimental): Open-label 2 mg baricitinib administered orally once daily (QD) to participants who randomized to placebo in the originating study (JAIW).
  Interventions: Drug: Baricitinib
- Baricitinib 1-mg/Baricitinib 2-mg (Experimental): Open-label 2 mg baricitinib administered orally QD to participants who randomized to 1 mg baricitinib in the originating study (JAIW).
  Interventions: Drug: Baricitinib
- Baricitinib 2-mg/Baricitinib 2-mg (Experimental): Open-label 2 mg baricitinib administered orally QD to participants who randomized to 2 mg baricitinib in the originating study (JAIW).
  Interventions: Drug: Baricitinib
- Baricitinib 2-mg Open-Label Addendum (Experimental): Participants were directly enrolled to receive open-label 2 mg baricitinib orally QD.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104

SUMMARY:
This open-label study will evaluate the long-term efficacy and safety of baricitinib in adult participants with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Have participated in Study JAIW (NCT03435081), and meet specific completion requirements for that study, and do not meet any of the following Exclusions:

* Have significant uncontrolled cerebro-cardiovascular (e.g., myocardial infarction [MI], unstable angina, unstable arterial hypertension, severe heart failure, or cerebrovascular accident), respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neuropsychiatric disorders, or abnormal laboratory values that developed during a previous baricitinib study that, in the opinion of the investigator, pose an unacceptable risk to the participant if investigational product continues to be administered.
* Have a known hypersensitivity to baricitinib or any component of this investigational product.
* Had investigational product permanently discontinued at any time during a previous baricitinib study, except for participants who had investigational product discontinued during originating study because of rescue with an oral systemic AD therapy (e.g., corticosteroid, cyclosporine, methotrexate).
* Had temporary investigational product interruption continue at the final study visit of a previous baricitinib study and, in the opinion of the investigator, this poses an unacceptable risk for the participant's participation in the study.
* Pregnant or breastfeeding

OR

• Have not participated in a Study JAIW (NCT03435081) and satisfy the following criteria:

Inclusion Criteria:

* Have a diagnosis of atopic dermatitis (AD) at least 12 months before screening.
* Have moderate to severe AD, including all of the following:

  * EASI score ≥16
  * IGA score of ≥3
  * 10%- 50% BSA involvement
* Have had inadequate response or intolerance to existing topical (applied to the skin) medications within 6 months preceding screening.
* Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments)
* Agree to use emollients daily.

Exclusion Criteria:

* Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus), or a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections.
* A history of eczema herpeticum within 12 months, and/or a history of 2 or more episodes of eczema herpeticum in the past.
* Participants who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics.
* Have any serious illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
* Have been treated with the following therapies:

  * monoclonal antibody for less than 5 half-lives before randomization
  * received prior treatment with any oral Janus kinase (JAK) inhibitor less than 4 weeks before randomization
  * received any parenteral corticosteroid administered by intramuscular or intravenous injection within 6 weeks of planned randomization or are anticipated to require parenteral injection of corticosteroids during the study
  * have had an intra-articular corticosteroid injection within 6 weeks of planned randomization
  * probenecid at the time of randomization that cannot be discontinued for the duration of the study
* Have high blood pressure characterized by a repeated systolic blood pressure >160 millimeters of mercury (mm Hg) or diastolic blood pressure >100 mm Hg.
* Have had major surgery within the past eight weeks or are planning major surgery during the study.
* Have experienced any of the following within 12 weeks of screening: myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of venous thromboembolic event (VTE), or are considered at high risk for VTE.
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, lymphoproliferative disease or neuropsychiatric disorders or any other serious and/or unstable illness.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection including herpes zoster, tuberculosis.
* Have specific laboratory abnormalities.
* Have received certain treatments that are contraindicated.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (74):
- United States (53):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johnson Dermatology, Fort Smith, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Keck School of Medicine University of Southern California, Los Angeles, California
  - Wallace Medical Group, Inc., Los Angeles, California
  - University of California Davis-Dermatology, Sacramento, California
  - Medical Center For Clinical Research, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Care Access Research-Walnut Creek, Walnut Creek, California
  - GWU/Medical Faculty Associates, Washington D.C., District of Columbia
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Olympian Clinical Research, Largo, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Riverchase Dermatology and Cosmetic Surgery, Pembroke Pines, Florida
  - University of South Florida, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Dermatologic Surgery Specialists, PC, Macon, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Advanced Clinical Research LLC, Meridian, Idaho
  - Northwestern University, Chicago, Illinois
  - University Dermatology, Darien, Illinois
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Forefront Research, Louisville, Kentucky
  - Dermatology and Skin Cancer Specialists, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Central Dermatology PC, St Louis, Missouri
  - Skin Specialists, P.C, Omaha, Nebraska
  - Icahn Sch of Med at Mt. Sinai, New York, New York
  - DermResearchCenter of New York, Inc, Stony Brook, New York
  - Bexley Dermatology Research, Bexley, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Wright State Univ School of Medicine, Fairborn, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - The Pennsylvania Centre for Dermatology, LLC, Exton, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Bellaire Dermatology, Bellaire, Texas
  - Modern Research Associates, Dallas, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - University of Utah MidValley Dematology, Murray, Utah
  - MultiCare Good Samaritan Hospital, Tacoma, Washington
- Canada (17):
  - Kirk Barber Research, Calgary, Alberta
  - Beacon Dermatology, Calgary, Alberta
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Simcoderm Medical & Surgical Dermatology Centre, Barrie, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Allergy Research Canada Inc., Niagara Falls, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Centre de Recherche Dermatologique de Quebec Metropolitain, Québec, Quebec
- Puerto Rico (4):
  - Dr. Samuel Sanchez PSC, Caguas, PR
  - Office of Dr. Alma M. Cruz, Carolina, PR
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - GCM Medical Group, PSC - Hato Rey Site, San Juan, PR

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Wollenberg A, Kircik L, Simpson E, Brinker D, Katoh N, Rueda MJ, Issa M, Yang F, Feely M, Alexis A. Pooled Analysis of Baricitinib Tolerability in Patients With Atopic Dermatitis in Relation to Acne, Headache, and Gastrointestinal Events From 8 Clinical Trials. Dermatitis. 2023 Jul-Aug;34(4):308-314. doi: 10.1089/derm.2022.0027. Epub 2023 Feb 6. PMID 36749121
- [Derived] King B, Maari C, Lain E, Silverberg JI, Issa M, Holzwarth K, Brinker D, Cardillo T, Nunes FP, Simpson EL. Extended Safety Analysis of Baricitinib 2 mg in Adult Patients with Atopic Dermatitis: An Integrated Analysis from Eight Randomized Clinical Trials. Am J Clin Dermatol. 2021 May;22(3):395-405. doi: 10.1007/s40257-021-00602-x. Epub 2021 Apr 7. PMID 33826132
- See also: A Study of Baricitinib (LY3009104) in Participants With Moderate to Severe Atopic Dermatitis — https://trials.lillytrialguide.com/en-US/trial/11hI0LRhfAAIAAa2qKq0ok

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants (nonresponder/partial responder: completed at least 16 weeks of treatment; responder: completed the full treatment period) from originating study JAIW (NCT03435081) enrolled into Open-label Treatment Period of JAIX [lasting from Week 0 (baseline through Week 200) or early termination visit]. Participants enrolled directly into Protocol Addendum I4V-MC-JAIX (2) without first completing at least 16 weeks of treatment in originating study JAIW.
Period: Overall Study
Arm/Group | Placebo/Baricitinib 2-milligram (mg) | Baricitinib 1-mg/Baricitinib 2-mg | Baricitinib 2-mg/Baricitinib 2-mg | Baricitinib 2-mg Open-Label Addendum
Started | 117 | 119 | 108 | 30
Received at Least One Dose of Study Drug | 117 | 119 | 108 | 30
Completed | 0 | 1 | 0 | 0
Not Completed | 117 | 118 | 108 | 30
Not completed — Adverse Event | 6 | 5 | 3 | 0
Not completed — Lack of Efficacy | 34 | 52 | 37 | 2
Not completed — Death | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 16 | 4 | 12 | 3
Not completed — Sponsor Decision | 38 | 31 | 35 | 18
Not completed — Withdrawal by Subject | 19 | 21 | 18 | 7
Not completed — Physician Decision | 3 | 2 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all participants who received at least one dose of study drug.
Groups:
- Placebo/Baricitinib 2-mg: Open-label 2 mg baricitinib administered orally QD to participants who randomized to placebo in the originating study (JAIW).
- Total: Total of all reporting groups
Arm/Group | Placebo/Baricitinib 2-mg | Baricitinib 1-mg/Baricitinib 2-mg | Baricitinib 2-mg/Baricitinib 2-mg | Baricitinib 2-mg Open-Label Addendum | Total
Number analyzed (Participants) | 117 | 119 | 108 | 30 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.90 (16.87) | 40.70 (16.86) | 39.30 (15.05) | 43.80 (17.67) | 40.30 (16.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 60 | 57 | 16 | 188
  Male | 62 | 59 | 51 | 14 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 13 | 19 | 10 | 59
  Not Hispanic or Latino | 97 | 105 | 87 | 20 | 309
  Unknown or Not Reported | 3 | 1 | 2 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 0 | 6
  Asian | 27 | 24 | 19 | 4 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 20 | 15 | 22 | 4 | 61
  White | 61 | 72 | 60 | 22 | 215
  More than one race | 6 | 5 | 4 | 0 | 15
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 36 | 38 | 31 | 0 | 105
  United States | 81 | 81 | 77 | 30 | 269

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI75)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
  The results were analyzed using non-responder imputation (NRI). All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as EASI75.
Time Frame: Week 16
Population: mITT population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Baricitinib 2-mg | Baricitinib 1-mg/Baricitinib 2-mg | Baricitinib 2-mg/Baricitinib 2-mg | Baricitinib 2-mg Open-Label Addendum
Number analyzed (Participants) | 117 | 119 | 108 | 30
percentage of participants | 59.0 | 40.3 | 45.4 | 50.0

2. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
  The results were analyzed using NRI. All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as IGA 0/1.
Time Frame: Week 16
Population: mITT population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Baricitinib 2-mg | Baricitinib 1-mg/Baricitinib 2-mg | Baricitinib 2-mg/Baricitinib 2-mg | Baricitinib 2-mg Open-Label Addendum
Number analyzed (Participants) | 117 | 119 | 108 | 30
percentage of participants | 44.4 | 18.5 | 29.6 | 40.0

3. Secondary Outcome: Percentage of Participants Achieving a Body Surface Area (BSA) of ≤3%
Description: The BSA affected by AD will be assessed for 4 separate body regions: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. BSA was calculated using the participant's palm using the 1% rule, 1 palm was equivalent to 1% with estimates of the number of palms it takes to cover the affected AD area. Maximum number of palms were 10 palms for head and neck (10%), 20 palms for upper extremities (20%), 30 palms for trunk, including axilla and groin (30%), 40 palms for lower extremities, including buttocks (40%). Percent of BSA for a body region was calculated as = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA of all 4 body regions ranges from 0% to 100 % with higher values representing greater severity of AD.
Time Frame: Week 16
Population: mITT population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Baricitinib 2-mg | Baricitinib 1-mg/Baricitinib 2-mg | Baricitinib 2-mg/Baricitinib 2-mg | Baricitinib 2-mg Open-Label Addendum
Number analyzed (Participants) | 117 | 119 | 108 | 30
percentage of participants | 39.3 | 21.8 | 35.2 | 43.3

4. Secondary Outcome: Percentage of Participants Achieving a ≥4-Point Improvement in Itch Numeric Rating Scale (NRS)
Description: The NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
Time Frame: Week 16
Population: mITT population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Baricitinib 2-mg | Baricitinib 1-mg/Baricitinib 2-mg | Baricitinib 2-mg/Baricitinib 2-mg | Baricitinib 2-mg Open-Label Addendum
Number analyzed (Participants) | 117 | 119 | 108 | 30
percentage of participants | 41.9 | 29.4 | 30.6 | 26.7

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up to 204 Weeks)
Description: All participants who received at least one dose of study drug and who did not discontinue from the study for the reason "Lost to Follow-up" at the first postbaseline visit in study.
Arm/Group | Placebo/Baricitinib 2-mg | Baricitinib 1-mg/Baricitinib 2-mg | Baricitinib 2-mg/Baricitinib 2-mg | Baricitinib 2-mg Open-Label Addendum
All-Cause Mortality (participants affected / at risk) | 0/117 | 2/119 | 0/108 | 0/29
Serious Adverse Events (participants affected / at risk) | 8/117 | 8/119 | 10/108 | 0/29
Other Adverse Events (participants affected / at risk) | 35/117 | 22/119 | 28/108 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Baricitinib 2-mg (N=117) | Baricitinib 1-mg/Baricitinib 2-mg (N=119) | Baricitinib 2-mg/Baricitinib 2-mg (N=108) | Baricitinib 2-mg Open-Label Addendum (N=29)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Graft infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer helicobacter (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cutaneous t-cell lymphoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Baricitinib 2-mg (N=117) | Baricitinib 1-mg/Baricitinib 2-mg (N=119) | Baricitinib 2-mg/Baricitinib 2-mg (N=108) | Baricitinib 2-mg Open-Label Addendum (N=29)
Covid-19 (Infections and infestations) | 9 (9) | 3 (3) | 5 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (14) | 9 (9) | 7 (7) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (13) | 8 (10) | 11 (15) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (14) | 6 (6) | 7 (9) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated before completion, due to lack of alignment during regulatory negotiations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: JAIX 05 Protocol (c).pdf (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT03559270/Prot_000.pdf
  • Study Protocol: JAIX 05 Protocol Addenda (2) (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT03559270/Prot_001.pdf
  • Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT03559270/SAP_002.pdf